CLINICAL TRIAL: NCT00347243
Title: Wavefront Analisys and Contrast Sensitivity of Spherical and Aspherical
Brief Title: Wavefront Analisys and Contrast Sensitivity of Spherical and Aspherical Intraocular Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP012/06
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-03

CONDITIONS: Cataract; Pseudophakia
MeSH Terms: conditions — Cataract; Pseudophakia | interventions — Phacoemulsification; Cataract Extraction

INTERVENTIONS:
Procedure: phacoemulsification (cataract surgery)

SUMMARY:
Purpose:To compare visual performance, total and high order wavefront aberrations (coma, spherical aberration and other terms) and contrast sensitivity in eyes implanted with one monofocal aspheric intraocular lens (IOL) and two spherical IOLs (SofPort AO, Soflex,AcrySof®IQ (40 eyes), AcrySof®Natural and AMO®Sensar)

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral visually significant senile cataract, corneal astigmatism less than 2.0 diopters and potential acuity meter (PAM) better than 0.2 LogMar

Exclusion Criteria:

* any other ocular diseases, such as corneal opacities or irregularity, dry eye, amblyopia, anisometropia, glaucoma, retinal abnormalities, surgical complications, IOL tilt, decentration (estimated by retro illumination and digital photo) greater than 0.4mm13 or loss of follow-up

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Schor, MD, Study Director — UNIFESP - EPM
Locations (1):
- Federal University of Sao paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Altmann GE. Wavefront-customized intraocular lenses. Curr Opin Ophthalmol. 2004 Aug;15(4):358-64. doi: 10.1097/00055735-200408000-00013. PMID 15232477